CLINICAL TRIAL: NCT03412864
Title: Post Marketing Surveillance on Safety and Effectiveness Evaluation of INVOSSA K Inj.
Brief Title: A Post Marketing Surveillance Study of INVOSSA K Inj.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kolon Life Science (Industry)
Responsible Party: Sponsor
Other Study IDs: KS-INVOSSA-PMS
Record Dates: First submitted 2018-01-19; First posted 2018-01-29 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis
Keywords: chondrocyte cells; osteoarthritis; gene therapy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is post-marketing surveillance of Invossa K injection in patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients over 19 years
2. Patients who diagnosed with osteoarthritis will plan to INVOSSA K Inj. injection and suitable for following criteria :

   - Moderate knee osteoarthritis (Kellgren & Lawrence grade 3) with persistent symptoms (pain, etc.) in spite of conservative therapy (medication, physical therapy, etc.) for more than 3 months
3. Patients (or substitute) who is provided all information regarding participation of this PMS signed the informed consent form

Exclusion Criteria:

1. Pregnant or breastfeeding female
2. Patients who have administered corticosteroid before INVOSSA K Inj. injection within the past 30 days
3. Patients who have severe disease such as heart, liver, kidney disease or other severe complications
4. Patients who rheumatoid arthritis, gouty arthritis, autoimmune disease associated arthritis except for osteoarthritis
5. Patients with a medical history of allergic diseases or patients with a medical history of anaphylactic reactions (including patients with a history of hypersensitivity reactions to the components of this drug, including dimethylsulfoxide (DMSO), mannitol, dextran 40 or bovine proteins)
6. Patients who have been treated with injections to the target knee within the past three months or patients with a past history of surgery, including arthroscope, within the past six months
7. Patients currently with leukemia or malignant tumors such as osteochondroma, chondroblastoma, cartilaginous mucinous fibrous tumor, chondroma and chondrosarcoma, which may be exacerbated by administration of INVOSSA-K inj. or patients with a history thereof
8. Patients with Kellgran & Lawrence grade 4 osteoarthritis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients over 19 years with osteoarthritis
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2023-07-11 (Estimated); Study Completion 2023-07-11 (Estimated)

PRIMARY OUTCOMES:
AEs (Adverse Events) | 0 month(visit 1), 1 month(visit 2) and 6 Months(visit 3)
  Changes of incidence rate in AEs

SECONDARY OUTCOMES:
100 mm VAS (Visual Analog Scale) | 0 month(visit 1), 1 month(visit 2) and 6 Months(visit 3)
  Changes of 100 mm VAS at each visit (Scale : 0~100, 0 : No pain, 100 : Worst imaginable pain)
Physical examination (Knee joint swelling) | 0 month(visit 1), 1 month(visit 2) and 6 Months(visit 3)
  Changes of Knee joint swelling at each visit
Physical examination (Tenderness) | 0 month(visit 1), 1 month(visit 2) and 6 Months(visit 3)
  Changes of tenderness at each visit
Physical examination (ROM) | 0 month(visit 1), 1 month(visit 2) and 6 Months(visit 3)
  Changes of ROM(Range Of Motion) at each visit
General efficacy evaluation | 6 Months(visit 3)
  General efficacy evaluation was assessed by following 4 criteria. (Improved, Not changed, Worsened, Unassessable)

CONTACTS AND LOCATIONS:
Overall Officials: Oog Jin Shon, MD, PhD., Principal Investigator — Yeungnam University Hospital
Locations (1):
- Yeungnam University Hospital, Daegu, Gyeongsangbuk-do, South Korea